CLINICAL TRIAL: NCT06750523
Title: Getting Bone Health Right From the Start: Innovative Technology and New Mechanims of Mother-fetus Cross Talk for Osteopenia and Osteporosis Prevention
Brief Title: Advancing Early Bone Health: New Frontiers for Osteoporosis Prevention
Acronym: REMS-BONE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Principal Investigator, Serafina Perrone, Professor, PhD, MD, University of Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ID SIRER 5484; PNRR-MAD-2022-12376819 (Other Grant/Funding Number: NEXTGENERATIONEU, Ministry of University and Research (MUR))
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Low-Risk Pregnant Women at Full-Term Gestation; Healthy Fetal Population; Healthy Neonatal Population
Keywords: Bone mineral Density; Fetus; Newborns; Children; Osteoporosis; Environment; Oxidative stress; Endocrine disruptors
MeSH Terms: conditions — Osteoporosis | interventions — Cordocentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mother and infants at term of physiologically gestation (<37 weeks) (Experimental): Assessment of bone mineral density (BMD) of the femur in the mother and fetus at term gestational age, and subsequently in the newborns at 48 hours after birth, at 1 month, at 3 months, at 6 months, and at 12 months of life, using REMS technology.
  Interventions: Diagnostic Test: Cord blood sampling; Diagnostic Test: urine sampling; Behavioral: Life style questionnaire

INTERVENTIONS:
Diagnostic Test: Cord blood sampling — A cord blood sample will be taken at birth for analysis of oxidative stress markers, endocrine disruptors, and microRNAs.
Diagnostic Test: urine sampling — At one month of age, urine samples will be collected from newborns to analyze oxidative stress markers and endocrine disruptors.
Behavioral: Life style questionnaire — At the time of enrollment, mothers will complete a specialized questionnaire designed to assess potential exposure to endocrine disruptors (EDCs) through diet, clothing, and the use of cosmetics and detergents.

SUMMARY:
All factors that influence the peak bone mass achieved at skeletal maturity are important in determining an individual's risk of developing osteoporosis later in life. Bone health begins with maternal health and nutrition, which influence skeletal mass and bone density in utero. The mechanisms underlying the effect of the intrauterine environment on bone health are currently unknown, but certainly include 'fetal programming' of oxidative stress and endocrine systems, as these influence skeletal growth and development later in life.

For the prevention of bone health, the challenges rely 1) in the need for new technology and software specific and applicable to the fetus and newborn; 2) in establishing the effect of environmental contaminants, in particular endocrine disruptors, oxidative stress and subsequent epigenetic changes in mothers and subsequently on the fetus, newborn and infant.

DETAILED DESCRIPTION:
Maximising bone mass during skeletal growth has become the goal of primary prevention of osteopenia and osteoporosis. Any factor that might influence the peak bone mass attained during skeletal maturation is important in determining an individual's risk of developing osteoporosis later in life. Bone health begins with maternal health and nutrition, which influence skeletal mass and bone density in the foetus. The acquisition of peak bone mass is also genetically influenced by both parents. To date, there is some evidence that the risk of osteoporosis in later life may be determined by environmental exposures during intrauterine or early postnatal life. The mechanisms underlying the long-term effects of the intrauterine environment on bone health are currently unknown, but certainly include "fetal programming" of oxidative stress and endocrine systems that influence skeletal growth and development in utero and after birth.

Osteopenia is increasingly diagnosed in low birth weight infants. Intrauterine growth restriction (IUGR) further increases the risk of obesity and metabolic syndrome, conditions that significantly compromise bone quality. Recent studies have highlighted the central role of microRNAs (miRNAs) in bone growth and mineralisation, alongside peptides such as irisin and HMGB-1. These peptides are involved in glucose metabolism and the regulation of adipose and muscle tissue and have recently been linked to bone metabolism. MicroRNAs and long non-coding RNAs (lncRNAs) have gained attention for their ability to regulate gene expression post-transcriptionally, providing epigenetic modifications that influence growth plate and bone development. It remains unclear how maternal nutritional factors affect fetal bone mineral density (BMD) or how variations in fetal BMD may influence birth outcomes, such as spontaneous clavicle or skull fractures during operative delivery, and long-term bone mineralisation.

These findings highlight the importance of assessing skeletal status during the perinatal period. Early identification of conditions that affect bone mass or mineralisation and ongoing monitoring of bone development are essential to improve outcomes.

Radiofrequency echographic multi-spectrometry (REMS) technology has demonstrated its utility in the assessment of BMD in pregnant women. While few studies have investigated the use of transmission ultrasound to assess bone status in neonates, REMS technology shows great promise. Its advantages include the absence of ionising radiation, ease of use and, most importantly, the potential to conduct longitudinal studies of REMS patterns from the intrauterine period into the first year of life.

This innovative approach offers new opportunities to understand the maternal-fetal factors that influence bone health and to develop strategies to optimise bone development from the earliest stages of life.

The aims of the present study are A) To determine the feasibility of using REMS as a precise and innovative technology to assess the skeletal status of fetuses, neonates and children.

B) To assess how maternal REMS patterns and her anthropometric and gestational data influence REMS parameters in the fetus, newborn and during the first year of life.

C) To elucidate the relationships between early exposure to endocrine disrupters, oxidative stress and maternal diet as part of the in utero exposome and later body composition and bone health.

ELIGIBILITY:
Inclusion Criteria:

* term infants from low-risk pregnancy
* (37-42 weeks gestational age)
* Single pregnancy
* Absence of current or previous maternal diseases that could potentially interfere with bone metabolism (e.g., thyroid, kidney, liver disease)
* Absence of motor disability of the mother
* No previous history of recent, previous bone fractures or traumatic fractures (in the mother)
* No intake of vitamin D or other medications during pregnancy
* Maternal age >18 years
* No diagnosis of osteopenia or osteoporosis according to the criteria of the Italian Society for Osteoporosis, Mineral Metabolism and Bone Diseases (SIOMMMS)

Exclusion Criteria:

* preterm infants
* Infants hospitalized since birth for special conditions
* infants with metabolic disorders
* infants with genetic syndromes

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | >37 and <42 weeks; 48 hours; 1, 3, 6, and 12 months
  The novel application of REMS technology in the fetal and neonatal population requires the construction of a reference database. Data from the first 100 enrolled fetuses will form the basis of this database, and the same approach will apply to newborns, with the initial 100 cases corresponding to the same fetal cohort. Echographic acquisitions of fetuses and newborns, obtained using REMS devices, will be anonymized and transferred to the subcontractor, who will adapt REMS configurations for pediatric use. This adaptation will enable the identification of target bone structures and provide densitometric outputs.
  BMD values will be calculated for each age group, and from the first 100 cases, mean and standard deviation will be derived to construct a 6-point BMD reference curve, comprising fetuses (>37 and <42 weeks) and newborns (48 hours, 1, 3, 6, and 12 months). Z-scores will be used to assess bone growth, and separate gender-specific curves will be developed.
MicroRNA assay on umbilical cord blood | at birth
  By TaqMan Advanced miRNA assays (Applied Biosystems) miRNAs will be quantified and normalized using hsa-miR-16-5p (Assay ID: 477860_mir) as endogenous control. Real-Time qRT-PCR will be used for the specific candidate miRNAs: miR-199a-5p, miR-140, miR-335-5p, mir-503-5p, miR-494-3p, mir-369-3p, mir-379-5p, as it has been recently shown that they vary in relationship to GH status, and are related to growth response.
Endocrine disruptors (EDCs) on umbilical cord blood at birth. | at birth
  Thirteen different EDCs are assayed, namely: Di(2-ethylhexyl) phthalate and its oxidised metabolites (MEHP, 6-OH-MEHP, 5-carboxy-MEPP, 5-oxo MEHP, 5-OH-MEHP), Bisphenol (BP) A, BPS, BPF, polyciclic aromatic hydrocarbons, polychorodibenzophuranes and polichorodibenzo-p-dioxins, perfluoro-alchilic substances, gliphosate, and its main metabolite, parabens (methyl-, ethyl-, propyl-, butyl- esters of 4-Hydroxybenzoic acid), piretroid insecticides,heavy metals (Pb, Cr).
Endocrine disruptors (EDCs) on urine at 1 months of age. | 1 month
  Thirteen different EDCs are assayed, namely: Di(2-ethylhexyl) phthalate and its oxidised metabolites (MEHP, 6-OH-MEHP, 5-carboxy-MEPP, 5-oxo MEHP, 5-OH-MEHP), Bisphenol (BP) A, BPS, BPF, polyciclic aromatic hydrocarbons, polychorodibenzophuranes and polichorodibenzo-p-dioxins, perfluoro-alchilic substances, gliphosate, and its main metabolite, parabens (methyl-, ethyl-, propyl-, butyl- esters of 4-Hydroxybenzoic acid), piretroid insecticides,heavy metals (Pb, Cr).
Oxidative stress (OS) profile | at birth, 1 month
  Oxidative stress (OS) profile will be evaluated by biomarkers of oxidative protein damage (Advanced Oxidation Protein Products, AOPP) and lipid peroxidation (Isoprostanes, IsoPs, malondialdehyde, MDA).
Oxidative stress (OS) molecules | at birth, 1 month
  Non-enzymatic antioxidant molecules (vitamin E; glutathione, GSH, and ascorbic acid, AA) and enzymatic antioxidant molecules (superoxide dismutase, SOD, catalase, CAT, and glutathione peroxidase, GPx) will be evaluated by highly specific and sensitive methods, such as high resolution liquid chromatography (HPLC), and gas chromatography interfaced mass spectrometry (GC-MS).
Lipid mediators involved in oxidative stress | at birth, 1 month
  The ELISA test will be used for the investigation of lipid metabolism and will evaluate specialised pro-resolving lipid mediators (Resolvin D1).
Standard biochemical tests | at birth, 1 month
  calcium, phosphorus, alkaline phosphatase, PTH, vitamin D (25 OH), and IGF-I
Exposure to endocrine disruptors (EDCs) related to diet, clothing and the use of cosmetics and detergents. | at the enrollment
  The questionnaire is an adaptation of the questionnaire drafted and already used as part of two previous projects "Phthalates and bisphenol A biomonitoring in Italianmother-childpairs: link between exposure and juvenile diseases' (LIFE PERSUADED) LIFE13 ENV/IT/000482; and 'Mother and infants dyads: lowering the impact of endocrine disrupting chemicals in milk for a healthy life2 (LIFE MILCH-LIFE18 ENV/EN/000460).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliero Universitaria "Gaetano Martino" di Messina, Messina, ME
  - Azienda Ospedaliero-Universitaria di Parma, Parma

REFERENCES:
- [Background] Heaney RP. BMD: the problem. Osteoporos Int. 2005 Sep;16(9):1013-5. doi: 10.1007/s00198-005-1855-y. Epub 2005 Mar 18. No abstract available. PMID 15776218
- [Background] Godfrey K, Walker-Bone K, Robinson S, Taylor P, Shore S, Wheeler T, Cooper C. Neonatal bone mass: influence of parental birthweight, maternal smoking, body composition, and activity during pregnancy. J Bone Miner Res. 2001 Sep;16(9):1694-703. doi: 10.1359/jbmr.2001.16.9.1694. PMID 11547840
- [Background] Lanham SA, Roberts C, Perry MJ, Cooper C, Oreffo RO. Intrauterine programming of bone. Part 2: alteration of skeletal structure. Osteoporos Int. 2008 Feb;19(2):157-67. doi: 10.1007/s00198-007-0448-3. Epub 2007 Aug 18. PMID 17704965
- [Background] Dirkes RK, Welly RJ, Mao J, Kinkade J, Vieira-Potter VJ, Rosenfeld CS, Bruzina PS. Gestational and lactational exposure to BPA, but not BPS, negatively impacts trabecular microarchitecture and cortical geometry in adult male offspring. Bone Rep. 2021 Nov 3;15:101147. doi: 10.1016/j.bonr.2021.101147. eCollection 2021 Dec. PMID 34820485
- [Background] Papaioannou G. miRNAs in Bone Development. Curr Genomics. 2015 Dec;16(6):427-34. doi: 10.2174/1389202916666150817202425. PMID 27019617
- [Background] Bocheva G, Boyadjieva N. Epigenetic regulation of fetal bone development and placental transfer of nutrients: progress for osteoporosis. Interdiscip Toxicol. 2011 Dec;4(4):167-72. doi: 10.2478/v10102-011-0026-6. PMID 22319250
- [Background] Holroyd C, Harvey N, Dennison E, Cooper C. Epigenetic influences in the developmental origins of osteoporosis. Osteoporos Int. 2012 Feb;23(2):401-10. doi: 10.1007/s00198-011-1671-5. Epub 2011 Jun 9. PMID 21656266
- [Background] Zhang L, Tang Y, Zhu X, Tu T, Sui L, Han Q, Yu L, Meng S, Zheng L, Valverde P, Tang J, Murray D, Zhou X, Drissi H, Dard MM, Tu Q, Chen J. Overexpression of MiR-335-5p Promotes Bone Formation and Regeneration in Mice. J Bone Miner Res. 2017 Dec;32(12):2466-2475. doi: 10.1002/jbmr.3230. Epub 2017 Aug 28. PMID 28846804
- [Background] Perrone S, Santacroce A, Picardi A, Buonocore G. Fetal programming and early identification of newborns at high risk of free radical-mediated diseases. World J Clin Pediatr. 2016 May 8;5(2):172-81. doi: 10.5409/wjcp.v5.i2.172. eCollection 2016 May 8. PMID 27170927
- [Background] Street ME, Bernasconi S. Endocrine-Disrupting Chemicals in Human Fetal Growth. Int J Mol Sci. 2020 Feb 20;21(4):1430. doi: 10.3390/ijms21041430. PMID 32093249
- [Background] Predieri B, Alves CAD, Iughetti L. New insights on the effects of endocrine-disrupting chemicals on children. J Pediatr (Rio J). 2022 Mar-Apr;98 Suppl 1(Suppl 1):S73-S85. doi: 10.1016/j.jped.2021.11.003. Epub 2021 Dec 15. PMID 34921754
- [Background] Degennaro VA, Brandi ML, Cagninelli G, Casciaro S, Ciardo D, Conversano F, Di Pasquo E, Gonnelli S, Lombardi FA, Pisani P, Ghi T. First assessment of bone mineral density in healthy pregnant women by means of Radiofrequency Echographic Multi Spectrometry (REMS) technology. Eur J Obstet Gynecol Reprod Biol. 2021 Aug;263:44-49. doi: 10.1016/j.ejogrb.2021.06.014. Epub 2021 Jun 15. PMID 34167032
- [Background] Basu S, Michaelsson K, Olofsson H, Johansson S, Melhus H. Association between oxidative stress and bone mineral density. Biochem Biophys Res Commun. 2001 Oct 19;288(1):275-9. doi: 10.1006/bbrc.2001.5747. PMID 11594785
- [Background] Wang X, Liang T, Zhu Y, Qiu J, Qiu X, Lian C, Gao B, Peng Y, Liang A, Zhou H, Yang X, Liao Z, Li Y, Xu C, Su P, Huang D. Melatonin prevents bone destruction in mice with retinoic acid-induced osteoporosis. Mol Med. 2019 Aug 28;25(1):43. doi: 10.1186/s10020-019-0107-0. PMID 31462213
- [Background] Perrone S, Laschi E, Buonocore G. Oxidative stress biomarkers in the perinatal period: Diagnostic and prognostic value. Semin Fetal Neonatal Med. 2020 Apr;25(2):101087. doi: 10.1016/j.siny.2020.101087. Epub 2020 Jan 23. PMID 32008959